CLINICAL TRIAL: NCT06694883
Title: Research on the Biological Basis of "Disease-Syndrome-Formula" in the Critical State of "Remission-Recurrence" of Ulcerative Colitis (Joint Application A)
Brief Title: Critical State of "Remission-Recurrence" of Ulcerative Colitis
Acronym: CSRRUC
Status: Recruiting | Type: Observational
Sponsor: Beijing Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Shengsheng Zhang, Principal Investigator, Beijing Hospital of Traditional Chinese Medicine
Other Study IDs: 82341235
Record Dates: First submitted 2024-11-03; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood,urine,stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ulcerative colitis in remission period

SUMMARY:
This study will recruit 100 patients with ulcerative colitis in remission for a 6-month non intervention follow-up observation. During the study, their conditions will be recorded truthfully, including general information, disease-related symptoms and signs, inflammatory bowel disease questionnaire, anxiety self-assessment scale, depression self-assessment scale, etc., every month. Collect blood, urine, and stool samples from patients every month for examination. Follow up for each subject until their condition recurs.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the criteria based on the clinical characteristics of ulcerative colitis patients in the "remission recurrence" critical state, combined with clinical symptoms, are diagnosed with ulcerative colitis through imaging, endoscopy, laboratory, and histopathological examinations;
* Patients with comprehensive laboratory testing indicators.

Exclusion Criteria:

* Patients with incomplete case information records;
* Patients who have not completed serological tests;
* Complications including intestinal obstruction, intestinal perforation, toxic megacolon, and severe local stenosis;
* Diagnosed or suspected patients with coexisting uncertain colitis, infectious or ischemic colitis;
* Patients with coexisting local or systemic infections, any malignant diseases, or autoimmune diseases;
* Merge primary diseases such as respiratory, circulatory, neurological, endocrine, and hematological disorders;
* Individuals at risk of developing cancer;
* regnant or lactating women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Visited the Digestive Department Outpatient Department of Beijing Hospital of Traditional Chinese Medicine
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
The recurrence rate of patients | The recurrence status of patients will be recorded during the 6-month follow-up period, and the recurrence rate will be calculated after all patients have completed the follow-up. It will take about 1 year to complete the entire process
  The recurrence rate of 100 follow-up patients was counted at the end of the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Shengsheng Zhang, Doctor, Principal Investigator — Beijing Hospital of Traditional Chinese Medicine
Locations (1):
- Beijing Hospital of Traditional Chinese Medicine, Capital Medical University, Dongcheng, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fukuda T, Naganuma M, Sugimoto S, Nanki K, Mizuno S, Mutaguchi M, Nakazato Y, Inoue N, Ogata H, Iwao Y, Kanai T. The risk factor of clinical relapse in ulcerative colitis patients with low dose 5-aminosalicylic acid as maintenance therapy: A report from the IBD registry. PLoS One. 2017 Nov 6;12(11):e0187737. doi: 10.1371/journal.pone.0187737. eCollection 2017. PMID 29108025
- [Background] Gordon GL, Zakko S, Murthy U, Sedghi S, Pruitt R, Barrett AC, Bortey E, Paterson C, Forbes WP, Lichtenstein GR. Once-daily Mesalamine Formulation for Maintenance of Remission in Ulcerative Colitis: A Randomized, Placebo-controlled Clinical Trial. J Clin Gastroenterol. 2016 Apr;50(4):318-25. doi: 10.1097/MCG.0000000000000414. PMID 26368296
- [Background] Segal JP, LeBlanc JF, Hart AL. Ulcerative colitis: an update. Clin Med (Lond). 2021 Mar;21(2):135-139. doi: 10.7861/clinmed.2021-0080. PMID 33762374